CLINICAL TRIAL: NCT03882164
Title: Use of Tacrolimus Blood-bile Ratio for the Detection of Early Liver Failure After Liver Transplantation
Brief Title: Blood-Bile Ratio Tacrolimus After Liver Transplantation
Acronym: BBRT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Dr. Marco Maria Pascale, Resident, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: PoliclinicoUAG-LTU
Record Dates: First submitted 2019-03-17; First posted 2019-03-20 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Liver Transplant; Complications; Immunosuppression; Transplant Failure; Transplant; Complication, Rejection
Keywords: Liver transplant;; Immunosuppression;; Transplant rejection;
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Biospecimen Retention: Samples Without DNA — Blood; Bile
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Rejection: Patient undergone liver transplant with diagnosis of rejection within 10 days
  Interventions: Diagnostic Test: Blood-Bile Ratio of Tacrolimus
- No-Rejection: Patient undergone liver transplant wothout diagnosis of rejection within 10 days

INTERVENTIONS:
Diagnostic Test: Blood-Bile Ratio of Tacrolimus — Diagnosis of early transplanted liver dysfunction to adjust Tacrolimus dose adminstered
  Groups: Rejection

SUMMARY:
Tacrolimus is the most widely used immunosuppressive drug in the prevention of rejection after solid organ transplantation. Pharmacokinetic studies in healthy volunteers and in transplanted patients have shown that this molecule is rapidly absorbed after oral administration (maximum plasma concentration after 1-2 hours), is found in the circulation bound mainly to erythrocytes and, after being metabolized by CYP3A4, is eliminated through the bile. The importance of the tacrolimus blood dosage is now widely recognized for detecting the immunosuppressive capacity reached in the individual patient or the eventual overdose of the drug. In the use of Tacrolimus after Liver Transplantation, however, it is interesting to note that the biochemical pathway for metabolism and excretion of the drug is present in the transplanted organ, the main object of immunological and functional surveillance. The excretory capacity of Tacrolimus by the liver through the bile, therefore, could be a useful tool for recognizing the early liver failure from a functional point of view, before the onset of hepatoecrosis.

DETAILED DESCRIPTION:
Prospective monocentric randomized study comparing two parallel groups:

liver transplanted patients with early (10 POD) organ rejection (experimental arm); liver transplanted patients without early (10 POD) organ rejection (control arm) Primary Objective: Evaluation of a correlation between the reduction of Tacrolimus biliary excretion and the early liver failure Primary Endpoint: Increase of Tacrolimus blood-bile ratio measured before the onset of laboratory hepatonecrosis Secondary Objective: Analysis of the cause of any drug-related toxicity Secondary Endpoint: correlation study between drug dosage and biliary excretion level in case of blood overdose or clinical evidence of pharmacological toxicity

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* History of recent liver transplant (less than 10 days)
* Placement of kehr tube in the biliary tract during liver transplant
* Immunosuppressive therapy with Tacrolimus
* Functioning of kehr tube

Exclusion Criteria:

* Age - Age ≥18 years
* History of liver transplant for more than 10 days
* Liver transplant without positioning of kehr tube
* Immunosuppressive therapy with a drug different from Tacrolimus
* No functioning of kehr tube18 years
* History of liver transplant for more than 10 days
* Liver transplant without positioning of kehr tube
* Immunosuppressive therapy with a drug different from Tacrolimus
* No functioning of kehr tube

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergone liver transplant with positioning of Kehr tube
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Analysis of early liver rejection | 10 days
  Evaluation of early liver rejection throught creation of a Tacrolimus blood-bile ratio

SECONDARY OUTCOMES:
Analysis of Tacrolimus toxicity | 10 days
  Evaluation of Tacrolimus toxicity throught blood dosage of the drug

CONTACTS AND LOCATIONS:
Locations (1):
- Marco Maria Pascale, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No